CLINICAL TRIAL: NCT03998592
Title: Phase I Clinical Trial for Assessment of Safety and Immunogenicity of a Synthetic Vaccine Against Streptococcus Pyogenes in Healthy Volunteers
Brief Title: Clinical Trial to Assess Safety and Immunogenicity of a Synthetic Vaccine Against Streptococcus Pyogenes
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Agreement between interested partied ended
Sponsor: Butantan Institute (Other Government)
Collaborators: InCor - Instituto do Coração - HCFMUSP. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EGA-01-IB
Record Dates: First submitted 2019-06-24; First posted 2019-06-26 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Rheumatic Fever
Keywords: vaccine; peptide; Streptococcus pyogenes
MeSH Terms: conditions — Rheumatic Fever

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Low-dose vaccine (Experimental)
  Interventions: Biological: Streptococcus pyogenes vaccine (50 µg)
- Mid-dose vaccine (Experimental)
  Interventions: Biological: Streptococcus pyogenes vaccine (100 µg)
- High-dose vaccine (Experimental)
  Interventions: Biological: Streptococcus pyogenes vaccine (200 µg)
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Streptococcus pyogenes vaccine (50 µg) — Vaccine containing 50 µg of StreptInCor synthetic peptide and Aluminium Hydroxide as adjuvant
  Arms: Low-dose vaccine
Biological: Streptococcus pyogenes vaccine (100 µg) — Vaccine containing 100 µg of StreptInCor synthetic peptide and Aluminium Hydroxide as adjuvant
  Arms: Mid-dose vaccine
Biological: Streptococcus pyogenes vaccine (200 µg) — Vaccine containing 200 µg of StreptInCor synthetic peptide and Aluminium Hydroxide as adjuvant
  Arms: High-dose vaccine
Other: Placebo — Placebo without active component
  Arms: Placebo

SUMMARY:
This is a double-blind, randomized, placebo-controlled phase I clinical trial with dose-escalation of a synthetic vaccine against Streptococcus pyogenes. The active component of this vaccine candidate is a synthetic polypeptide named StreptInCor designed to elicit humoral and cell-mediated immune responses. The vaccine will be formulated with Aluminium hydroxide in three different doses of StreptInCor (50 µg, 100µg, 200 µg). The proposed vaccination schedule is three doses (0, 1, 6 months). The doses will be escalated for the next group after safety review.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers, both sex, aging 18 to 45 years;
* Availability for all procedures during the study period;
* Provide free informed consent to join the study

Exclusion Criteria:

* Diagnosis of concomitant infections or diseases that might affect immunity, including active HIV infection, hepatitis B, hepatitis C, diabetes mellitus, neoplasias, and autoimmune diseases;
* Previous or current diagnosis or family antecedent of rheumatic fever, chorea, obsessive-compulsive disorder or glomerulonephritis;
* Previous or current diagnosis of cardiac disease;
* Severe asma or Chronic obstructive pulmonary disease (COPD);
* Abnormal neurological clinical assessment, particularly chorea;
* Use of treatments that might affect the immunity in the last four weeks, including immunomodulators, corticosteroids (only systemic use equal or longer than two weeks), or antineoplastic agents;
* Use of treatments that might affect heart valves in the latest four weeks, including fenfluramine e dexfenfluramine;
* Kidney failure determined by creatinine clearance lower than 45 ml/min/1,73m²;
* History of intolerance or allergy to any component of investigational products, including antigen or adjuvant;
* Presence of abnormalities in heart valves or heart anatomy defined by echocardiogram;
* Electrocardiogram disturbances;
* Presence of cross-reactive antibodies against human tissues (heart, kidney, cartilage, brain) in screening tests;
* Evidence or suspicion of recent infection due to S. pyogenes assessed by clinical symptoms and negative rapid test for Streptococcus;
* Pregnancy, breastfeeding mother or intention to became pregnant during the study period;
* Any other condition that might affect the study process according to the investigators.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-05 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Solicited and unsolicited adverse reactions | Six months after last dose
  Frequency of solicited and unsolicited adverse reactions
Immune response to vaccine | Six months after last dose
  Rate of seroconversion for vaccine epitopes

CONTACTS AND LOCATIONS:
Overall Officials: Luiza Guilherme, PhD, Study Chair — InCor Heart Institute; Roney O Sampaio, MD, PhD, Principal Investigator — InCor Heart Institute

IPD SHARING:
Plan to Share IPD: No